CLINICAL TRIAL: NCT00257946
Title: Prospective Randomized Trial Comparing Type of Material in Repair of Congenital Diaphragmatic Hernia
Brief Title: Type of Material in Repair of Congenital Diaphragmatic Hernia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: poor accrual
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Shawn St. Peter, Associate Professor, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0510128
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Congenital Diaphragmatic Hernia
Keywords: Diaphragm; Hernia; Congenital
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital; Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Repair of CDH w/SIS Gold
Procedure: Repair of CDH w/Alloderm

SUMMARY:
The objective of this study is to evaluate the use of 2 different types of biosynthetic material for the repair of congenital diaphragmatic hernia. The research question is: what is the best material for repairing large congenital diaphragmatic hernias? The primary outcome variable is recurrence.

DETAILED DESCRIPTION:
At birth, the estimated gestational age and birth weight will be recorded, as well as the presence and type of other congenital anomalies.

Prior to operation, the length of time from birth to repair will be recorded. To determine the severity of physiologic compromise, the need and type of ventilator support as well as the need and length of ECMO support will be recorded. The amount of time between ECMO discontinuation and repair will be recorded. The respiratory support required at the time of operation will be recorded.

At operation, the size of the defect will be measured and recorded. The location (right versus left) will be recorded and special notation will be recorded regarding any areas where no diaphragmatic rim is present. The operative time and charges will be recorded.

After the operation, the length of ventilator support, time to feeds, hospital stay, and hospital charges will be recorded. Post-operative complications such as bleeding complications, pneumonia, sepsis, gastroesophageal reflux, early recurrence and bowel obstruction will be recorded. Future operations and type of procedure will be recorded. If future operations in the abdomen are required, the amount and severity of intraperitoneal adhesions will be noted and recorded. Mortality will be recorded.

After discharge, commensurate with standard current clinical practice, all patients will receive a follow-up appointment with a chest x-ray at 6 months and 1 year of life. After this time, follow-up appointments will be made each year for the first 5 years of life and imaging will be obtained on the basis of symptoms. Any further follow-up will be as needed for symptoms. Oxygen requirements, findings at follow-up and future hospitalization will be recorded, particularly looking at the presence or absence of hernia recurrence. The study will mature and effectively close when all subjects have reached 5 year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Infants admitted to the neonatal intensive care unit with a diagnosis of congenital diaphragmatic hernia as proven by chest x-ray showing enteric contents in the thoracic cavity will be considered. Those who have birth weight equal to or over 2.2 kilograms and who are at or beyond 34 weeks gestation at the time of birth who survive until an operation can be performed will be considered. At operation, the patients with posterolateral diaphragmatic defects (Bockdalek Hernia) large enough to require placement of a patch to recreate the diaphragm will be included in the study.

Exclusion Criteria:

* Children diagnosed outside of the neonatal period will not be considered. Patients with the less common anteromedial or substernal defect (Morgagni Hernia) will not be included in the study as their physiology and rate of recurrence are incomparable to common posterolateral, Bockdalek Hernia.

Those patients under 2.2 kilograms and less than 34 weeks gestation have poor lung maturity to compound their inherent difficulty with pulmonary parenchymal hypoplasia and pulmonary vasculature hypertension making their chances of survival extremely low. Further compounding their dismal circumstance, they are not candidates for salvage extracorporeal membrane oxygenation (ECMO). Therefore, they will not be candidates for the study.

The rare case requiring repair of the hernia while on ECMO support will not be included due to the fact that this population has a very poor survival secondary to irreversible pulmonary hypertension. Further, the operation is performed while the patient is anticoagulated with heparin which is fraught with operative and post-operative bleeding.

Max Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50
Dates: Start 2005-12; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Recurrence of Diaphragmatic Hernia

SECONDARY OUTCOMES:
Bowel Obstruction
Ventilatory days
Ventilatory status at follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Shawn D St. Peter, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States